CLINICAL TRIAL: NCT03539133
Title: Systemic Organ Communication in STEMI
Acronym: SYSTEMI
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 17-018
Record Dates: First submitted 2018-05-03; First posted 2018-05-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: STEMI; infarction; coronary artery disease; comorbidities; diabetes; anemia
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Infarction; Coronary Artery Disease; Diabetes Mellitus; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — prospectively defined blood sampling protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collection of clinical data — prospectively and systematically collection of clinical research data from STEMI patients

SUMMARY:
Despite progress in pre-hospital care, ambulance logistics, pharmacotherapy and PPCI techniques, ST-segment elevation myocardial infarction (STEMI) continues to confer a substantial burden of morbidity and mortality.

Within the STEMI population, there is a spectrum of higher and lower risk patients. The aim of this cohort study is to collect prospectively and systematically clinical research data from STEMI patients. This cohort study is an open-end observational study to identify master switches in myocardial ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from STEMI

Exclusion Criteria:

* < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from STEMI
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Left-ventricular function | 6 months
  * LV-EF < 40% at 6 months
  * Δ LV-EF ≥ 5% between day 5 of hospitalization and 6 months
Left-ventricular remodeling | 6 months
  Δ LVEDV ≥ 20% or Δ LVESV ≥ 15% between day 5 of hospitalization and 6 months
Myocardial texture | on day 5 of hospitalization and 6 months
  * Infarct/Scar size > 17.9% or MVO (yes) or IMH (yes) on day 5 of hospitalization or at 6 months
  * remote zone ΔECV between day 5 of hospitalization and 6 months
Patency rate | 6 months
  Coronary patency rate

SECONDARY OUTCOMES:
All cause mortaltiy | 12 months
  All cause mortaltiy
MACCE | 12 months
  cardiovascular death, non-fatal stroke or myocardial infarction
Re-Hospitalisation due to heart failure | 12 months
  Re-Hospitalisation due to heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jung, MD, PhD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

REFERENCES:
- [Derived] Benkhoff M, Alde K, Ehreiser V, Dahlmanns J, Metzen D, Haurand JM, Duse DA, Jung C, Kelm M, Petzold T, Polzin A. Thromboinflammation is associated with clinical outcome after ST-elevation myocardial infarction. Blood Adv. 2024 Nov 12;8(21):5581-5589. doi: 10.1182/bloodadvances.2024014273. PMID 39226457
- [Derived] Bonner F, Jung C, Polzin A, Erkens R, Dannenberg L, Ipek R, Kaldirim M, Cramer M, Wischmann P, Zaharia OP, Meyer C, Flogel U, Levkau B, Godecke A, Fischer J, Klocker N, Kruger M, Roden M, Kelm M. SYSTEMI - systemic organ communication in STEMI: design and rationale of a cohort study of patients with ST-segment elevation myocardial infarction. BMC Cardiovasc Disord. 2023 May 3;23(1):232. doi: 10.1186/s12872-023-03210-1. PMID 37138228